CLINICAL TRIAL: NCT06461663
Title: An Interventional, Post-Market Study to Evaluate the Performance of a Custom-made Medical Device, "Breast Cancer Locator (BCL)" System, in Breast-conserving Surgery (BCS)
Brief Title: CairnSurgical Breast Cancer Locator (BCL) Post-Market Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CairnSurgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-BCL-EU2021
Record Dates: First submitted 2023-01-09; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All subjects will undergo breast conserving surgery with the BCL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment with BCL (Experimental): Subjects will undergo breast conserving surgery with the Breast Cancer Locator (BCL)
  Interventions: Device: Breast Cancer Locator Guided Breast Conserving Surgery

INTERVENTIONS:
Device: Breast Cancer Locator Guided Breast Conserving Surgery — Subjects will undergo a contrast-enhanced supine MRI and two marks will be placed on the breast. The MRI images will be transmitted to the sponsor, and the images will be used to build a BCL using 3D printing. Investigators will be provided with a 3D image of the cancer in the breast. Investigators will use a BCL (a patient-specific, plastic, bra-like form that is placed on the breast and allows the investigator to mark the edges of the tumor on the skin and to place wires inside the breast which define the center of the cancer and the tumor edges. The surgeon will then attempt to surgically remove all the tissue inside the wires used to define the tumor edges.

SUMMARY:
This interventional, post-market, multicenter clinical investigation is designed to evaluate the performance of a custom-made medical device, "the Breast Cancer Locator (BCL)" in Subjects with non-palpable breast cancer, in Europe.

DETAILED DESCRIPTION:
The aim of this interventional, post-market, multicenter clinical investigation is to evaluate the performance of a custom-made medical device, the Breast Cancer Locator (BCL) system, in subjects with non-palpable breast cancer. The study will be conducted in European countries. To evaluate the performance of BCL in reducing the positive margin rate, the proportion of patients with positive margins after partial mastectomy with the BCL will be obtained.

Each Subject, after signing an Informed Consent Form (ICF), will enter into a screening phase, during which several assessments (e.g., demographics, medical history, evaluation of available prone MRI and core biopsy pathological results) will be conducted.

At visit 1, the Subject will undergo supine MRI, from which a 3D breast image and BCL will be made.

At visit 2, the patient will undergo Breast Conserving Surgery (BCS) using the BCL system. On the same day, the specimen volume will be determined. The excised specimen will be sent to the pathological lab for analysis. The results, including the positive margin rate (PMR) and specimen mammogram, will be obtained within 14 days.

At visit 3, follow-up assessments (including physical examination, and adverse event review) will be performed.

At the End Of Study visit, adverse events will be assessed and patients will be asked to express their satisfaction with the BREAST-Q.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed
* Female Aged ≥ 18 years at the time of the signature of ICF
* Histologic diagnosis of IBC or DCIS
* Tumor excision that will require localization because it cannot be definitively defined by palpation
* The tumor is unifocal; possible satellite lesions < 2 cm from primary are eligible
* The tumor enhances and is greater than or equal to 5mm on prone breast MRI imaging
* Subject and surgeon agree to perform BCS
* Willingness to follow all study procedures, including attending all site visits, tests and examinations.

Exclusion Criteria:

* Absolute contraindication to MRI, including presence of implanted electrical device (e.g., pacemaker or neurostimulator), aneurysm clip, or metallic foreign body in or near eyes
* Severe claustrophobia
* Contraindication to use of gadolinium-based intravenous contrast, including life-threatening allergy
* Uncontrolled cardiac, renal, or pulmonary disease
* Uncontrolled systemic disease (e.g., lupus erythematosus or scleroderma)
* Compromised renal function including chronic, severe kidney disease (GFR < 30 ml/min/1.73m2), or acute kidney injury
* Pregnancy or breast-feeding
* Subjects who have received or plan to receive neoadjuvant chemotherapy
* Sternal notch to nipple distance of > 32 cm as measured in a sitting or standing position
* Measurement of widest circumference around breasts and arms > 135 cm
* Known allergy to device components
* Multicentric tumors (additional tumors > 2 cm from primary)
* Infectious or inflammatory processes near the area of intervention
* Planned surgery with localization devices including WGL, intraoperative ultrasound guidance, radiofrequency emitting implants, magnetic seeds, radioactive seeds, and tissue inspection devices
* Simultaneous participation in an interventional study or participation in an interventional study in the last 1 month before study inclusion
* Known drug and/or alcohol abuse
* Mental incapacity that precludes adequate understanding or cooperation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Positive Margin Rate | Pathology results will from the index procedure be available within 14 days from the day of sample arrival at the pathological lab.
  To evaluate the performance of BCL in reducing the positive margin rate, the proportion of patients with positive margins after partial mastectomy with the BCL will be obtained.

SECONDARY OUTCOMES:
Specimen volume | Results will be obtained the same day of surgery.
  To calculate the specimen volume after BCL guided partial mastectomy, the water displacement method (WDM) will be used.
Surgeon's Perception | Results will be obtained prior to subject discharge after the study procedure (within approximately 2 days after surgery)
  To evaluate the surgeon's perception of the BCL system, a survey asking them if they strongly disagree, somewhat disagree, are undecided, somewhat agree, or strongly agree that the BCL made tumor localization easier, was easy to use, made tumor excision easier, and would be recommended by them, will be used.
Adverse events | From supine MRI 10-40 days prior to surgery through 6 weeks +/- 7 days post surgery
  To evaluate the safety and tolerability of BCL, adverse events will be reported, including frequency, maximum intensity, relation to study treatment, seriousness, action taken, and outcome. Safety data will be handled descriptively.
Patient Satisfaction | 6 weeks +/- 7 days post surgery
  To evaluate the patient's satisfaction, the BREAST-Q patient-reported outcome measure will be used. Patient satisfaction scores range from 0-100, with a higher score meaning greater satisfaction or better quality of life (depending on the scale).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Barth, MD, Study Director — Cairn Surgical
Locations (5):
- Germany (2):
  - Agaplesion Markus Hospital, Frankfurt
  - Universitats Klinikum Heidelberg, Heidelberg
- Italy (2):
  - Humanitas Research Hospital, Milan
  - Ospdale Santa Chiara, Pisa
- Spital Zollikerberg, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to other researchers.